CLINICAL TRIAL: NCT04258358
Title: Evaluating the Community Areas of Sustainable Care and Dementia Excellence Model of Care
Acronym: CASCADE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unanticipated delays including those caused by COVID-19
Sponsor: Canterbury Christ Church University (Other)
Collaborators: Interreg (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: 2S02038
Record Dates: First submitted 2020-01-29; First posted 2020-02-06 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Dementia
Keywords: Dementia care; Community integrated care; Strengths-based approach; Technology; Person centered care
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Intervention Model Description: The factorial model examines the effect of using technology (telehealth) and learning and development resources on the cost of delivering dementia care and the well being of people living with dementia, family carers and staff delivering care.
  The learning and development resources hosted in an accessible repository will comprise three modular training modules at three different levels of healthcare professionals, carers and the public. The training modules include principles of CASCADE, person centred leadership and learning climate (giving and receiving feedback).
  Technology
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- People living with dementia intervention group (Experimental): Long term care and support are provided in a dementia care friendly environment with emphasis on 'the person's home'. Each resident's home carries a registered address to symbolise the person's home. Based on needs and strengths, people living with dementia and their families are supported to choose the technology to enable the person's independence plus developing new and maintaining existing skills. Examples of supportive and assistive technology include mobile devices, memory clocks, gas and flood detectors, sensor mats and global positioning system trackers or safe return ornaments. Routine care follows a holistic integrated health and social care plan tailored to the needs of the person living with dementia.
  Respite care provided in guesthouse facilities embody a similar approach only for a shorter period of time without assigning registered home addresses.
  Interventions: Other: CASCADE ways of working
- People living with dementia control group (No Intervention): People living with dementia in need of long-term rehabilitation or recovery for at least eight months; and people living with dementia in need of respite care for up to 14 days
  People living with dementia will continue to use standard care. Standard care in this respect constitutes usual health and social care or any other nationally acceptable form of therapy that people living with dementia would seek to use.

INTERVENTIONS:
Other: CASCADE ways of working — Technology, learning and development resources and nursing and therapeutic care are the key drivers for the CASCADE ways of working promoting community integrated dementia care and support to optimise safety and independence for people living with dementia.
  Other Names: Supportive care through CASCADE ways of working
  Arms: People living with dementia intervention group

SUMMARY:
The study evaluates the impact and cost effectiveness of community integrated dementia care. Some of the people living with dementia participating in the study will receive long term or respite care and support in the community tailored to CASCADE ways of working. Other people living with dementia participating in the study will continue to use standard care as usual. The terms 'CASCADE model of care' and 'CASCADE ways of working' are used here interchangeably as appropriate.

DETAILED DESCRIPTION:
The CASCADE ways of working draw on the person's strengths to optimize safety and independent living in their community. The ways of working incorporate learning and development for all stakeholders to enhance interactions with people living with dementia; use of technology to improve access to specialist care as well as safety in the community; and holistic care tailored to the needs of the person to improve and maintain well being. These elements work in tandem to enable people living with dementia to engage in meaningful leisure and activities of daily living.

The evaluation study aims to explore the benefits of the CASCADE model of care (ways of working) on service users (people with dementia and their caregivers), staff and service providers. The evaluation comprises elements of outcome and process evaluation. The outcome evaluation involves quantitative measures of health, well being and cost benefits while the process evaluation explores intervention implementation procedures to find out what worked and how it worked. The CASCADE model of care assumes that using the person's strengths to guide holistic personalized dementia care is a sustainable approach to safe meaningful independent living and improving public perceptions.

Investigators will use a quasi-experiment to assess quantifiable benefits (health and well being outcomes and cost benefits) of the CASCADE model for people with dementia. This means, investigators will compare two groups of people with dementia including one that will receive care under the CASCADE model (intervention group) and the second group will not. The anticipation is that comparing the two groups will make benefits of people receiving care under the CASCADE ways of working more observable. Participants will not be allocated randomly to the study arms because service use will be dependent on assessed need for referrals and need and affordability for self-referred users. This implies there is no opportunity to randomize participants to either the intervention or control groups. Time point measures will include pre-intervention (T0), and two follow up points (T1 and T2).

It is anticipated that 160 people living with dementia will take part in the study (respite intervention group n= 50; respite control group n=50; long term care intervention group n= 30; long term care control group n= 30). Other participants will include family or informal carers (n= 20) and staff delivering care (n=70).

The residential mode of the intervention will minimize cases of missing data. However, in the event of missing data, investigators will use Multiple Imputations Methods (MIM) if missing data are less than twenty percent (<20%). It is unlikely that data will be Missing Completely at Random (MCAR), but data Missing at Random will be assessed using appropriate statistical procedures such as analysis via the patterns command to determine patterns of missingness and their frequency and to examine variables predictive of missing data. Investigators will eliminate dropouts or noncompliance from analyses, if missing data are more than 20%. Similarly, if data are not Missing at Random, investigators will use last observation carried forward (LOCF) method particularly for participants in long term care to maintain the sample size and minimize confounding effects of noncompliance or attrition.

ELIGIBILITY:
Inclusion Criteria:

Specific inclusion criteria for long-term residents:

- The person needs long-term rehabilitation or recovery for at least eight months.

Specific inclusion criteria for guesthouse facilities

* The person needs emergency respite due to unforeseen circumstances
* In need of planned respite for example, due to informal carer's scheduled commitments
* The person needs short-term rehabilitation or recovery
* Using guesthouse with care facilities for a minimum of 14 days.

Exclusion Criteria:

* People with complex care needs that cannot be met at the project delivery sites during initial recruitment.
* People that will not consent to participate in the evaluation study.
* People living with dementia involved in other studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-05 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Quality Adjusted Life Years (QALYs) | 8 months
  The primary outcome will be Quality Adjusted Life Years (QALYs) for people living with dementia generated through the CASCADE ways of working. Health related quality of life will be measured using the EuroQol Group -Five Dimensions - Five-level scale (EQ-5D-5L). Results of EQ-5D-5L will be converted to utility values multiplied by the time spent in each state to generate QALYs. 1 QALY is equivalent to perfect health while less than perfect health carries a QALY between 0 and 1. A 0 QALY represents death. The higher the number of QALYs gained through the CASCADE model of care the better the health outcomes for people living with dementia.
Resource utilisation in dementia | 8 months
  A Resource Utilization in Dementia (RUD) scale will be used to assess use of hospital beds and other health and social care specialist services as well as informal carer's time and health. Less health specialists care used and low or no hospitalisation episodes in the intervention group compared to the control group implies higher cost benefits resulting from the CASCADE ways of working.

SECONDARY OUTCOMES:
Quality of life of people living with dementia | 8 months
  Investigators will measure changes on the quality of life of people living with dementia in the intervention group using the Quality of Life in Alzheimer's Disease (QOL-AD) scale. The maximum score obtainable on the13 items scale is 52 while the lowest score is 13. The higher the score the better the quality of life.
Quality of life of informal/ family carers | 8 months
  The Adult Carer Quality of Life (Ac-QoL) will be used to evaluate the quality of life of informal carers of people living with dementia in the intervention group. Scores on the Ac-QoL range from 0-120, higher scores showing better quality of life.

OTHER OUTCOMES:
Well being of staff delivering care | 8 months
  The Strain and Emotional Reaction in Dementia Care scale will be used to evaluate the impact of CASCADE ways of working on staff's well being. The scale comprises three domains assessing perceptions of behavior of people living with dementia evaluated on Likert scales.
  Positive attitude towards behavioural experiences, assessment of emotions and ease of handling challenges during care processes indicate greater wellbeing of staff delivering care and meaningful caring relationships.
Cost effectiveness | 8 months
  The cost of Quality Adjusted Life Years (QALYs) of people living with dementia in the intervention group will be compared with the control group to illustrate cost effectiveness of the CASCADE ways of working. Incremental Cost Effectiveness Ratio (ICER) will represent the additional cost per unit of QALY to indicate the trade-off between total cost and effectiveness of the CASCADE intervention compared to standard care.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Martin, Principal Investigator — Canterbury Christ Church University; Eleni Hatzidimitriadou, PhD, Study Chair — Canterbury Christ Church University
Locations (2):
- United Kingdom (2):
  - East Kent Hospitals University National Health Service Foundation Trust, Canterbury, Kent
  - Medway Community Healthcare, Rochester, Kent

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data underpinning results in publications, for example, data that underlie cost effectiveness of the intervention and health and wellbeing results for people living with dementia will be shared through publishing platforms. Individual participant datasets will be shared via a suitable public data repository. A description of the dataset shared and respective relationships will be included in the data repository.
  An evaluation study report will be made available through the Canterbury Christ Church University CASCADE project web page.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: It is anticipated the study protocol will be published in a suitable journal by December 2020. Individual participant data sets relating to the study will be made available via an appropriate data repository starting 6 months after formal publication of results.
  The evaluation study report will be available on Canterbury Christ Church University CASCADE project web page by April 2021.
Access Criteria: Anonymised data sets unpinning publications will be shared through the control measures of the publishing journals such as full access to subscribers